CLINICAL TRIAL: NCT03982485
Title: Neoadjuvant Apatinib Added to Weekly Paclitaxel and Cisplatin in Patient With Locally Advanced or Early Stage HER2 Negative Breast Cancer (APP) : a Open-label, Randomized, Controlled, Trial
Brief Title: Combination Neoadjuvant Chemotherapy With or Without Apatinib for HER2 Negative Breast Cancer
Acronym: APP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHPD005
Record Dates: First submitted 2019-04-10; First posted 2019-06-11 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: Apatinib; Neoadjuvant chemotherapy; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — apatinib; Paclitaxel; Cisplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Apatinib+Paclitaxel+Cisplatin
  Interventions: Drug: Apatinib; Drug: Paclitaxel; Drug: Cisplatin; Procedure: Surgery
- Arm II (Active Comparator): Paclitaxel+Cisplatin
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Procedure: Surgery

INTERVENTIONS:
Drug: Apatinib — Apatinib 250mg, Oral, day 2,3,4,5,6,7, every week
  Arms: Arm I
Drug: Paclitaxel — Paclitaxel 80mg/m2, Intravenous, day 1, 8, 15, 22, every 28 days for a cycle
Drug: Cisplatin — Cisplatin 25mg/m2, Intravenous, day 1, 8, 15, every 28 days for a cycle
Procedure: Surgery — Surgery

SUMMARY:
RATIONALE:

The combination of anti-angiogenic targeted therapy with neoadjuvant chemotherapy has been shown to further improve the pathologic response rate for HER2-negative breast cancer patients. Apatinib is a highly potent human vascular endothelial growth factor receptor 2 (VEGFR2) tyrosine kinase inhibitor that has been independently developed in China, and it can exert anti-angiogenic effects by inhibiting VEGFR2. It is unknown whether giving combination neoadjuvant chemotherapy together with apatinib is more effective in treating patients with nonmetastatic HER2-negative breast cancer.

PURPOSE:

To explore the efficacy and safety of apatinib added to weekly paclitaxel and cisplatin neoadjuvant therapy for HER-2 negative breast cancer patients

ELIGIBILITY:
Inclusion Criteria:

1. 18~70 year-old，Female
2. Patients with histologically confirmed primary invasive breast adenocarcinoma,cT2-4N0-3M0
3. ECOG 0-1
4. HER2-negative tumor in biopsy, defined as: Immunohistochemical (IHC) 0-1+ or IHC 2+ confirmed as FISH negative.
5. Adequate organ function

Exclusion Criteria:

1. Unwilling to use adequate contraceptive protection during the process of the study and for at least 8 weeks after the last dose of study drug.
2. Pregnant or breastfeeding patients
3. Metastatic or recurrent patients
4. Any evidence of sense or motor nerve disorders
5. Any concurrent malignancy other than breast cancer
6. Uncontrolled hypertension with hypotensive drugs therapy (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg). Patients with grade I or above myocardial ischemia or myocardial infarction or arrhythmia (including QT interval ≥ 440 ms) or cardiac insufficiency
7. Inability to swallow, gastrointestinal resection, chronic diarrhea and obstruction of the intestine, various factors which affect drug use and absorption
8. Coagulation disorders
9. Artery or venous thrombosis occurred within 6 months before the study begins
10. Have received prior treatment with a VEGFR TKI

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2031-03-29 (Estimated)

PRIMARY OUTCOMES:
Residual cancer burden (RCB 0-I rates） | Time of surgery
  RCB 0-I rates means RCB 0+I (good response) rates.
Pathologic Complete Response (pCR) of the Primary Tumor in the Breast | Time of surgery
  Percentage of patients absent of histologic evidence of invasive tumor cells in the surgical breast specimen.

SECONDARY OUTCOMES:
pCR in the Breast and Nodes | Time of surgery
  Percentage of patients absent of histologic evidence of invasive tumor cells in the surgical breast specimen and axillary lymph nodes.
Near pCR in the Breast | Time of surgery
  Percentage of patients with the residual breast lump Less than 10%
Clinical and imaging response | Time of surgery
  To determine the response rates of the breast tumor and axillary nodes based on physical examination and imaging tests. (sonography, mammography, or MRI) after treatment
Number of Participants With Drug Related Treatment Adverse Events | an average of 16 weeks
  Adverse events that occurred on or after initial treatment that were absent before treatment or worsened during the treatment period relative to the pretreatment state.
Neo-bioscore | Time of surgery
  The Neo-Bioscore staging points were determined for each patient based on information from the medical records according to the previously published work（Mittendorf EA, et al. The Neo-Bioscore Update for Staging Breast Cancer Treated With Neoadjuvant Chemotherapy: Incorporation of Prognostic Biologic Factors Into Staging After Treatment. JAMA Oncol. United States; 2016;2:929-36.）.
  Neo-Bioscore = Clinical stages score + Pathological stages score + Tumor marker score Clinical stage I =0, Clinical stage IIA =0, Clinical stage IIB =1, Clinical stage IIIA =1, Clinical stage IIIB =2, Clinical stage IIIC =2, Pathological stage 0 =0, Pathological stage I =0, Pathological stage IIA =1, Pathological stage IIB =1, Pathological l stage IIIA =1, Pathological stage IIIB =1, Pathological stage IIIC =2, Tumor marker ER negative=1 Tumor marker Grade3=1 Tumor marker ERBB2 negative=1
Disease-free Survival (DFS) | Measured through 5 years after study enrollment
  DFS is defined as the time period between registration and first event
Distant-disease- free survival (DDFS) | Measured through 5 years after study enrollment
  DDFS is defined as the time period between registration and first event
Overall survival (OS) | Measured through 5 years after study enrollment
  OS is defined as the time period between registration and first event

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Lu, MD, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China